CLINICAL TRIAL: NCT06410521
Title: Personalisation of Non-surgical Treatment in Peripheral Arterial Disease Using a Multicomponent Exercise Approach
Brief Title: Personalised Multicomponent Exercise Programme in Peripheral Arterial Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Trás-os-Montes and Alto Douro (Other)
Collaborators: Research Center in Sports Sciences, Health Sciences and Human Development (Other); Hospital Centre Hospitalar de Trás-os-Montes e Alto Douro (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PASSUS 2.0
Record Dates: First submitted 2024-05-07; First posted 2024-05-13 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Peripheral Arterial Disease; Intermittent Claudication
Keywords: Peripheral arterial disease; Supervised multicomponent exercise programme
MeSH Terms: conditions — Peripheral Arterial Disease; Intermittent Claudication | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: The study design will comprise two evaluation moments: initial evaluation (M0 - 0 week) and final evaluation (M1 - 12 weeks after). After M0 patients will be randomised into the intervention arm (experimental group) and comparator arm (usual care group). The intervention arm will perform supervised exercise (cardiovascular and resistance training) three times a week for 12 weeks and the comparator arm will receive information regarding standard lifestyle modification but without specific recommendations about the exercise programme.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Supervised multicomponent exercise (Experimental): Experimental arm will perform the supervised exercise programme three times a week, with each session taking approximately 60-80 minutes for a period of 12 weeks.
  Interventions: Behavioral: Exercise
- Usual care (Active Comparator): Active comparator arm will be advised to lifestyle modification and to perform regular walking for a period of 12 weeks.
  Interventions: Behavioral: Usual care

INTERVENTIONS:
Behavioral: Exercise — Patients randomised to the intervention arm will undergo non-consecutive training sessions three times a week for a period of 12 weeks. The training session is divided into an aerobic and a resistance training component, with a 5-min warm-up (stretching exercises) and a 5-min cool-down (stretching and relaxing exercises). The cardiovascular component will comprise a progressive exercise duration from 30 to 40 minutes, an exercise intensity promoting moderate to severe claudication pain between 8-12 minutes, with rest time until the pain disappears, and a personalised load progression manipulated based on the claudication pain level, reaching a total of 60 minutes of walking per session. The resistance training component will comprise dynamic muscle contraction exercises (Leg extension, unilateral hip extension, and standing calf raise), with a load progression from 50% of 1-estimated one repetition maximum (e-RM) to 80% of 1-eRM.
  Arms: Supervised multicomponent exercise
Behavioral: Usual care — Patients randomised to the active comparator arm will be advised about the importance of lifestyle modification (including general advice to increase walking but without specific recommendations about the exercise program) for a period of 12 weeks.
  Arms: Usual care

SUMMARY:
Peripheral arterial disease (PAD) is characterised as an atherosclerotic disease, most common in the lower limbs (aortoiliac, femoropopliteal, and infrapopliteal arterial segments), which causes a decrease in blood flow to the areas adjacent to and posterior to the affected area. Intermittent claudication (IC) is the most common symptom in this disease that appears with exertion and relieves with rest, causing fatigue, cramps, discomfort, or pain in the lower limbs due to limited blood flow to the affected muscles. Supervised physical exercise has emerged as the first line of intervention in improving the symptoms of intermittent claudication and disease progression, and in the last decade there has been an exponential increase in the use of wearable technologies to monitor dose-response. However, the approach used is still simplistic because it is not personalised. In other words, patients with similar diagnoses and symptoms get the same treatment, without personalising the stimulus according to their exercise responses and level of adaptation. With this in mind, this study aims to monitoring the real-time response of a multicomponent exercise programme (cardiovascular and resistance training) to personalise the dose-response, and use artificial intelligence models to gather and analyse vast amounts of data towards grouping/differentiating based on individual responses. The main hypothesis is that a supervised multicomponent exercise programme will improve the functional capacity of patients with PAD in a cluster personalised approach.

DETAILED DESCRIPTION:
Framework: Continuous monitoring of training allows for a better understanding and adjustment of the proposed objectives, based on the physiological responses provided. With the use of wearables increasing significantly and emerging as the main trend since 2016, near-infrared spectroscopy (NIRS) has been gaining emphasis as method for assessing muscle oxygen saturation (SmO2) and is an important tool in exercise monitoring. In the field of PAD, the use of NIRS is also fundamental as it allows the oxygen available in the muscle to be visualised in real time. NIRS technology makes it possible to observe the response to exercise in detail, in terms of deoxygenation and reoxygenation, which are essential analysis processes since PAD is characterised by oxygen insufficiency and the responses are highly individualised. In conjunction, the use of high-precision accelerometry (1600 Hz) helps to identify all the movements made by analysing the responses in the different axes. Based on the considerable gap in the literature regarding the effect of continuous monitoring and personalisation of the dose-response in this population, this study aims to assess the effect of a multicomponent cardiovascular and resistance training programme, personalised, and continuously monitored through heart rate (HR) and SmO2.

The experimental design comprises the following phases: i) programme design; ii) sample recruitment; iii) initial evaluation of the experimental group (Supervised exercise training) and the control group (Usual care) (M0 - 0 week); iv) personalisation of the exercise load; v) programme implementation; and vi) final evaluation of both groups (M1 - 12 weeks after).

Sample: Patients with PAD will be recruited at the Local Health Unit of Trás-os-Montes and Alto Douro, by the Angiology and Vascular Surgery Service. Participation in the study will be voluntary and written informed consent will be obtained from each patient. After the baseline assessments patient will be randomised to 1 of 2 groups, using a random number program with blocking to assure that the group sizes do not differ by >2.

Intervention: There will be two study arms: i) intervention arm - 12 weeks of supervised exercise (cardiovascular and resistance training) three times a week; and ii) comparator arm - a usual care group that will be instructed according to standard lifestyle modification but without specific recommendations about the exercise programme.

Power and sample size calculations: Power analysis performed in G*Power software (using ANOVA repeated measures within-between factors), version 3.1.9.7 (Institut für Experimentelle Psychologie, Düsseldorf, Germany) for an effect size of 0.25, an α of 0.05, and a power of 0.80 (1-ß) showed that 34 patients would be needed to achieve statistical significance. Considering the potential loss to follow-up, an attrition rate of 10% will be added to the calculated n, totalling 38 patients to be recruited.

Statistical analysis: Statistical analyses will be carried out using JASP software, version 0.18.1 (JASP Team, 2023) and the figures produced in GraphPad Prism software, version 8.0.1 (GraphPad Software, San Diego, California).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with clinically stable PAD;
* An ankle-brachial index (ABI) between 0.41-0.90 at rest in one or both lower limbs;
* Mild to moderate claudication, corresponding to Fontaine Stage IIa and IIb;
* A history of ambulatory leg pain;
* Ambulatory leg pain confirmed by treadmill test;
* Able to provide written consent.

Exclusion Criteria:

* Noncompressible, calcified, tibial arteries (resting ABI ≥ 1.4);
* Use of medication that could influence claudication (e.g. Cilostazol or Pentoxifylline) 3 months prior to investigation;
* Previous intervention (e.g. balloon angioplasty, stenting, bypass, exercise programme);
* Inability to walk on a treadmill at a speed of 3.2 km/h (2 mph);
* Participation in the past 3 months in a clinical trial or exercise program;
* Asymptomatic PAD determined from the medical history;
* Exercise limited by factors other diseases or conditions than intermittent claudication;
* Angina pectoris, congestive heart failure, chronic obstructive pulmonary disease, severe arthritis, or limb amputation.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-06-20 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Pain-free walking distance | Baseline and 12 weeks
  Distance until onset of claudication (in meters) will be measured in patients undergoing the graded treadmill exercise test (Gardner-Skinner protocol).
Maximum walking distance | Baseline and 12 weeks
  Walking distance until maximum claudication (in meters) will be measured in patients undergoing the graded treadmill exercise test (Gardner-Skinner protocol).
Percentage of muscle deoxygenation | Baseline and 12 weeks
  The percentage of muscle deoxygenation (in %) will be measured in patients undergoing the graded treadmill exercise test (Gardner-Skinner protocol).
Muscle reoxygenation time | Baseline and 12 weeks
  The muscle reoxygenation time (in seconds) will be measured in patients undergoing the graded treadmill exercise test (Gardner-Skinner protocol).

SECONDARY OUTCOMES:
Pain-free walking distance | Baseline and 12 weeks
  Distance until onset of claudication (in meters) will be measured in patients undergoing the 6-minute walk test.
Maximum walking distance | Baseline and 12 weeks
  Walking distance until maximum claudication (in meters) will be measured in patients undergoing the 6-minute walk test.
Percentage of muscle deoxygenation | Baseline and 12 weeks
  The percentage of muscle deoxygenation (in %) will be measured in patients undergoing the 6-minute walk test.
Muscle reoxygenation time | Baseline and 12 weeks
  The muscle reoxygenation time (in seconds) will be measured in patients undergoing the 6-minute walk test.
Lower limb muscle strength assessment | Baseline and 12 weeks
  The peak force (in kg) will be measured in patients using the hand-held dynamometry test.
Lower limb muscle power assessment | Baseline and 12 weeks
  The rate of force development (in kg/s) will be measured in patients using the hand-held dynamometry test.
Resting systolic blood pressure | Baseline and 12 weeks
  The resting systolic blood pressure (in mmHg) will be measured in patients after a 10-minute rest in a lying position.
Resting diastolic blood pressure | Baseline and 12 weeks
  The resting diastolic blood pressure (in mmHg) will be measured in patients after a 10-minute rest in a lying position.
Life quality | Baseline and 12 weeks
  The quality of life will be measured in patients using the 36-Item Short Form Survey that contains the domains of mental component and physical component.
Daily walking ability | Baseline and 12 weeks
  The daily walking will be measured in patients using the Walking Impairment Questionnaire that contains the domains of walking distance, walking speed and ability to climb stairs.
Fasting blood glucose | Baseline and 12 weeks
  The fasting blood glucose (in mg/dL) will be measured in patients using the fasting blood glucose test.
Sedentary behaviour | Baseline and 12 weeks
  The sedentary behaviour (in min/day) will be measured in patients over seven consecutive days.
Moderate-to-vigorous physical activity | Baseline and 12 weeks
  Moderate-to-vigorous physical activity (in min/day) will be measured in patients over seven consecutive days.

OTHER OUTCOMES:
Ankle-brachial index | Baseline and 12 weeks
  The ankle-brachial index (in a.u.) will be measured in patients after a 10-minutes rest in a lying position.
Body composition | Baseline and 12 weeks
  The body composition (the unit will depend on the derived-parameters evaluated) will be measured in patients in the orthostatic position according to guidelines.
Cross-sectional area of the gastrocnemius medialis muscle | Baseline and 12 weeks
  The cross-sectional area of the gastrocnemius medialis muscle of both lower limbs will be determined through an echographic evaluation.

CONTACTS AND LOCATIONS:
Overall Officials: Catarina Abrantes, Ph.D., Principal Investigator — University of Trás-os-Montes and Alto Douro, Vila Real, Portugal
Locations (3):
- Portugal (3):
  - Hospital Centre Hospitalar de Trás-os-Montes e Alto Douro, Vila Real
  - Research Centre in Sports Sciences, Health Sciences and Human Development, Vila Real
  - University of Trás-os-Montes and Alto Douro, Vila Real

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aboyans V, Ricco JB, Bartelink MEL, Bjorck M, Brodmann M, Cohnert T, Collet JP, Czerny M, De Carlo M, Debus S, Espinola-Klein C, Kahan T, Kownator S, Mazzolai L, Naylor AR, Roffi M, Rother J, Sprynger M, Tendera M, Tepe G, Venermo M, Vlachopoulos C, Desormais I; ESC Scientific Document Group. 2017 ESC Guidelines on the Diagnosis and Treatment of Peripheral Arterial Diseases, in collaboration with the European Society for Vascular Surgery (ESVS): Document covering atherosclerotic disease of extracranial carotid and vertebral, mesenteric, renal, upper and lower extremity arteriesEndorsed by: the European Stroke Organization (ESO)The Task Force for the Diagnosis and Treatment of Peripheral Arterial Diseases of the European Society of Cardiology (ESC) and of the European Society for Vascular Surgery (ESVS). Eur Heart J. 2018 Mar 1;39(9):763-816. doi: 10.1093/eurheartj/ehx095. No abstract available. PMID 28886620
- [Background] Baltrunas T, Mosenko V, Mackevicius A, Dambrauskas V, Asakiene I, Rucinskas K, Narmontas P. The use of near-infrared spectroscopy in the diagnosis of peripheral artery disease: A systematic review. Vascular. 2022 Aug;30(4):715-727. doi: 10.1177/17085381211025174. Epub 2021 Jun 10. PMID 34112030
- [Background] Cornelis N, Chatzinikolaou P, Buys R, Fourneau I, Claes J, Cornelissen V. The Use of Near Infrared Spectroscopy to Evaluate the Effect of Exercise on Peripheral Muscle Oxygenation in Patients with Lower Extremity Artery Disease: A Systematic Review. Eur J Vasc Endovasc Surg. 2021 May;61(5):837-847. doi: 10.1016/j.ejvs.2021.02.008. Epub 2021 Mar 30. PMID 33810977
- [Background] Nordanstig J, Behrendt CA, Bradbury AW, de Borst GJ, Fowkes F, Golledge J, Gottsater A, Hinchliffe RJ, Nikol S, Norgren L. Peripheral arterial disease (PAD) - A challenging manifestation of atherosclerosis. Prev Med. 2023 Jun;171:107489. doi: 10.1016/j.ypmed.2023.107489. Epub 2023 Apr 7. PMID 37031910
- [Background] Perrey S, Ferrari M. Muscle Oximetry in Sports Science: A Systematic Review. Sports Med. 2018 Mar;48(3):597-616. doi: 10.1007/s40279-017-0820-1. PMID 29177977